CLINICAL TRIAL: NCT04961060
Title: Drivers of Eosinophilic COPD Exacerbations
Acronym: DICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Maastricht University (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Maarten van den Berge, Principal Investigator, University Medical Center Groningen
Other Study IDs: NL75151.042.20
Record Dates: First submitted 2021-04-28; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: COPD Exacerbation; Eosinophilia
MeSH Terms: conditions — Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Eosinophilic exacerbation: COPD exacerbation associated with eosinophilia.
- Viral exacerbation: COPD exacerbation associated with viral infection.
- Bacterial exacerbation: COPD exacerbation associated bacterial infection.
- Pauci-inflammatory exacerbation: Pauci-inflammatory COPD exacerbation

SUMMARY:
Main objective: investigate gene expression differences in nasal epithelium and sputum between eosinophilic COPD exacerbations and other subtypes.

DETAILED DESCRIPTION:
Main objective: investigate gene expression differences in nasal epithelium and sputum between eosinophilic COPD exacerbations and other subtypes to better understand why some patients are more at risk for eosinophilic COPD exacerbations. Secondary objectives:

1. Investigate differences in microbiome composition and immunophenotyping profiles in peripheral blood per subtype.
2. Assess for clinical differences between all COPD exacerbation subtypes.
3. Assess if and how baseline meta-transcriptomics either in nasal epithelium or sputum and blood immunophenotyping can be utilized to predict COPD exacerbation subtype.
4. Determine if the microbiome in sputum and nasal epithelial material are comparable.
5. Determine if different subtypes of COPD exacerbations respond differently to standard treatment with oral prednisolone (40 mg daily) with or without antibiotics.
6. To evaluate if metabolic responses during recovery are different in patients with increased systemic inflammation compared to patients without systemic inflammation at exacerbation

ELIGIBILITY:
Inclusion Criteria:

1. COPD patient admitted to the hospital for an acute exacerbation of COPD
2. Physician diagnosed COPD according to the GOLD 2020 guidelines, including symptoms consistent with COPD, post-bronchodilator FEV1 < 80% predicted and FEV1/FVC < 70%.
3. Age > 40 years.
4. Smoker or ex-smoker, ≥ 10 pack years of smoking.

Exclusion Criteria:

1. Current asthma, or prior physician diagnosis of asthma without a symptom- free interval of at least 10 years before the age of 40.
2. Chronic use of prednisolone.
3. Use of systemic corticosteroids ≥4 days prior to hospital admission.
4. Necessity (upon hospitalization) for non-invasive ventilation or ICU admission.
5. Pneumonia at presentation documented by chest roentgenography.
6. Any other clinically relevant lung disease deemed to interfere with the concept of the study design.
7. Allergy to systemic corticosteroids or to antibiotics.
8. Females of childbearing potential without an efficient contraception unless they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH >40 mIU/mL or the use of one or more of the following acceptable methods of contraception:

   1. Surgical sterilization (e.g. bilateral tubal ligation, hysterectomy).
   2. Hormonal contraception (implantable, patch, oral, injectable).
   3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/suppository.
   4. Continuous abstinence
9. Pregnancy or lactation.
10. Known immunodeficiency.
11. Life expectancy less than 60 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the UMCG or MUMC for a COPD exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in gene expression profiles in sputum by RNA sequencing | At admission and after 6-8 weeks after discharge.
  Change in gene expression profiles in sputum between the four groups using RNA sequencing. The differences between the expression levels of transcripts (counts) will be analyzed.
Change in gene expression profiles in nasal epithelium by using RNA sequencing | At admission and after 6-8 weeks after discharge.
  Change in gene expression profilesin nasal epithelium between the four groups using RNA sequencing. The differences between the expression levels of transcripts (counts) will be analyzed.

SECONDARY OUTCOMES:
Microbiome composition in sputum by using RNA sequencing. | At admission, at day 5 of admission and 6-8 weeks after discharge.
  Differences in microbiome composition in sputum between the four groups by using RNA sequencing.
Phenotype blood cell population by flow cytometry. | At admission, at day 5 of admission and 6-8 weeks after discharge.
  Differences in blood cell population between the four groups as measured by flow cytometry.
Phenotypic analysis of the T cell compartment by staining of whole blood or isolated peripheral blood mononuclear cells using antibodies | At admission, at day 5 of admission and 6-8 weeks after discharge.
  Differences in the T cell compartment between the four groups by staining of whole blood or isolated peripheral blood mononuclear cells using antibodies.
Comparison of microbiome composition in sputum and nasal epithelial material by RNA sequencing. | At admission and 6-8 weeks after discharge.
  Measure microbiome composition in sputum and nasal epithelium by RNA sequencing. Compare them by the bacterial taxa which are significantly different between groups
Clinical differences between groups by the COPD Assessment Test (CAT). | Every day of hospital admission.
  Differences in number of participants per group with a high impact of COPD related symptoms as assessed by the CAT.
Clinical differences between groups by peak flow measurements. | Every day of hospital admission.
  Differences in number of participants per group with a low peak expiratory flow rate as measured by a handheld peak flow meter.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Maastricht, Maastricht, Limburg
  - Univesity Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Z, Singh R, Miller BE, Tal-Singer R, Van Horn S, Tomsho L, Mackay A, Allinson JP, Webb AJ, Brookes AJ, George LM, Barker B, Kolsum U, Donnelly LE, Belchamber K, Barnes PJ, Singh D, Brightling CE, Donaldson GC, Wedzicha JA, Brown JR; COPDMAP. Sputum microbiome temporal variability and dysbiosis in chronic obstructive pulmonary disease exacerbations: an analysis of the COPDMAP study. Thorax. 2018 Apr;73(4):331-338. doi: 10.1136/thoraxjnl-2017-210741. Epub 2017 Dec 21. PMID 29269441
- [Background] Bafadhel M, McKenna S, Terry S, Mistry V, Reid C, Haldar P, McCormick M, Haldar K, Kebadze T, Duvoix A, Lindblad K, Patel H, Rugman P, Dodson P, Jenkins M, Saunders M, Newbold P, Green RH, Venge P, Lomas DA, Barer MR, Johnston SL, Pavord ID, Brightling CE. Acute exacerbations of chronic obstructive pulmonary disease: identification of biologic clusters and their biomarkers. Am J Respir Crit Care Med. 2011 Sep 15;184(6):662-71. doi: 10.1164/rccm.201104-0597OC. PMID 21680942
- [Background] Mayhew D, Devos N, Lambert C, Brown JR, Clarke SC, Kim VL, Magid-Slav M, Miller BE, Ostridge KK, Patel R, Sathe G, Simola DF, Staples KJ, Sung R, Tal-Singer R, Tuck AC, Van Horn S, Weynants V, Williams NP, Devaster JM, Wilkinson TMA; AERIS Study Group. Longitudinal profiling of the lung microbiome in the AERIS study demonstrates repeatability of bacterial and eosinophilic COPD exacerbations. Thorax. 2018 May;73(5):422-430. doi: 10.1136/thoraxjnl-2017-210408. Epub 2018 Jan 31. PMID 29386298
- [Background] Imkamp K, Berg M, Vermeulen CJ, Heijink IH, Guryev V, Kerstjens HAM, Koppelman GH, van den Berge M, Faiz A. Nasal epithelium as a proxy for bronchial epithelium for smoking-induced gene expression and expression Quantitative Trait Loci. J Allergy Clin Immunol. 2018 Jul;142(1):314-317.e15. doi: 10.1016/j.jaci.2018.01.047. Epub 2018 Mar 6. No abstract available. PMID 29522853
- [Background] Boudewijn IM, Lan A, Faiz A, Cox CA, Brouwer S, Schokker S, Vroegop SJ, Nawijn MC, Woodruff PG, Christenson SA, Hagedoorn P, Frijlink HW, Choy DF, Brouwer U, Wisman M, Postma DS, Fingleton J, Beasley R, van den Berge M, Guryev V. Nasal gene expression changes with inhaled corticosteroid treatment in asthma. Allergy. 2020 Jan;75(1):191-194. doi: 10.1111/all.13952. Epub 2019 Jul 15. No abstract available. PMID 31230369
- [Background] Liesker JJ, Bathoorn E, Postma DS, Vonk JM, Timens W, Kerstjens HA. Sputum inflammation predicts exacerbations after cessation of inhaled corticosteroids in COPD. Respir Med. 2011 Dec;105(12):1853-60. doi: 10.1016/j.rmed.2011.07.002. Epub 2011 Jul 29. PMID 21802933
- [Background] Caramori G, Casolari P, Barczyk A, Durham AL, Di Stefano A, Adcock I. COPD immunopathology. Semin Immunopathol. 2016 Jul;38(4):497-515. doi: 10.1007/s00281-016-0561-5. Epub 2016 May 13. PMID 27178410
- [Background] Brusselle GG, Joos GF, Bracke KR. New insights into the immunology of chronic obstructive pulmonary disease. Lancet. 2011 Sep 10;378(9795):1015-26. doi: 10.1016/S0140-6736(11)60988-4. PMID 21907865
- [Background] Zhu J, Paul WE. Peripheral CD4+ T-cell differentiation regulated by networks of cytokines and transcription factors. Immunol Rev. 2010 Nov;238(1):247-62. doi: 10.1111/j.1600-065X.2010.00951.x. PMID 20969597
- [Background] Travers J, Rothenberg ME. Eosinophils in mucosal immune responses. Mucosal Immunol. 2015 May;8(3):464-75. doi: 10.1038/mi.2015.2. Epub 2015 Mar 25. PMID 25807184
- [Background] Aguirre-Gamboa R, Joosten I, Urbano PCM, van der Molen RG, van Rijssen E, van Cranenbroek B, Oosting M, Smeekens S, Jaeger M, Zorro M, Withoff S, van Herwaarden AE, Sweep FCGJ, Netea RT, Swertz MA, Franke L, Xavier RJ, Joosten LAB, Netea MG, Wijmenga C, Kumar V, Li Y, Koenen HJPM. Differential Effects of Environmental and Genetic Factors on T and B Cell Immune Traits. Cell Rep. 2016 Nov 22;17(9):2474-2487. doi: 10.1016/j.celrep.2016.10.053. Epub 2016 Nov 3. PMID 27818087
- [Background] Narendra DK, Hanania NA. Targeting IL-5 in COPD. Int J Chron Obstruct Pulmon Dis. 2019 May 16;14:1045-1051. doi: 10.2147/COPD.S155306. eCollection 2019. PMID 31190789
- [Background] Ditz B, Christenson S, Rossen J, Brightling C, Kerstjens HAM, van den Berge M, Faiz A. Sputum microbiome profiling in COPD: beyond singular pathogen detection. Thorax. 2020 Apr;75(4):338-344. doi: 10.1136/thoraxjnl-2019-214168. Epub 2020 Jan 29. PMID 31996401
- [Background] Gao P, Gibson PG, Zhang J, He X, Hao Y, Li P, Liu H. The safety of sputum induction in adults with acute exacerbation of COPD. Clin Respir J. 2013 Jan;7(1):101-9. doi: 10.1111/j.1752-699X.2012.00291.x. Epub 2012 Apr 23. PMID 22452898
- [Background] Pavord ID, Chanez P, Criner GJ, Kerstjens HAM, Korn S, Lugogo N, Martinot JB, Sagara H, Albers FC, Bradford ES, Harris SS, Mayer B, Rubin DB, Yancey SW, Sciurba FC. Mepolizumab for Eosinophilic Chronic Obstructive Pulmonary Disease. N Engl J Med. 2017 Oct 26;377(17):1613-1629. doi: 10.1056/NEJMoa1708208. Epub 2017 Sep 11. PMID 28893134
- [Background] Criner GJ, Celli BR, Brightling CE, Agusti A, Papi A, Singh D, Sin DD, Vogelmeier CF, Sciurba FC, Bafadhel M, Backer V, Kato M, Ramirez-Venegas A, Wei YF, Bjermer L, Shih VH, Jison M, O'Quinn S, Makulova N, Newbold P, Goldman M, Martin UJ; GALATHEA Study Investigators; TERRANOVA Study Investigators. Benralizumab for the Prevention of COPD Exacerbations. N Engl J Med. 2019 Sep 12;381(11):1023-1034. doi: 10.1056/NEJMoa1905248. Epub 2019 May 20. PMID 31112385
- [Background] Bi R, Liu P. Sample size calculation while controlling false discovery rate for differential expression analysis with RNA-sequencing experiments. BMC Bioinformatics. 2016 Mar 31;17:146. doi: 10.1186/s12859-016-0994-9. PMID 27029470
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Celli BR, Locantore N, Tal-Singer R, Riley J, Miller B, Vestbo J, Yates JC, Silverman EK, Owen CA, Divo M, Pinto-Plata V, Wouters EFM, Faner R, Agusti A; ECLIPSE Study Investigators. Emphysema and extrapulmonary tissue loss in COPD: a multi-organ loss of tissue phenotype. Eur Respir J. 2018 Feb 7;51(2):1702146. doi: 10.1183/13993003.02146-2017. Print 2018 Feb. PMID 29437944